CLINICAL TRIAL: NCT01264471
Title: Mechanisms of Mitochondrial Defects in Gulf War Syndrome
Status: Completed | Type: Observational
Sponsor: Medical Neurogenetics, LLC (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, John M. Shoffner, Medical Director, Medical Neurogenetics, LLC
Other Study IDs: H09378; GW080138 (Other Grant/Funding Number: Department of Defense CDMRP)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Gulf War Syndrome; Mitochondrial Disease
Keywords: Gulf War Syndrome; Gulf War Illness; Mitochondrial defects; Mitochondrial disorders; Persian Gulf Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome; Mitochondrial Diseases | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gulf War Syndrome patients: Gulf War veterans who have been diagnosed with Gulf War Syndrome.
  Interventions: Procedure: Skin biopsy; Procedure: Blood Collection

INTERVENTIONS:
Procedure: Skin biopsy — A small skin sample will be obtained from the patients arm which is approximately the size of the top of a thumbtack (a small circle no more than a 1/4 inch across)
  Other Names: skin sample
Procedure: Blood Collection — Approximately 45ml or 3 tablespoons for blood will be drawn from a vein in the patient's forearm.
  Other Names: phlebotomy; blood draw

SUMMARY:
The purpose of the study is to investigate possible causes for Gulf War Syndrome. Gulf War Syndrome is associated with increased incidences of amyotrophic lateral sclerosis (Lou Gehrig's Disease), pain syndromes, muscle complaints that include fatigue and myalgias (muscle pain), as well as other neurological symptoms. Abnormalities in the part of the cell known as mitochondria have been delineated in Gulf War Syndrome. Mitochondria are the "power plants" of the body. Mitochondria take the food you eat and break the food down into a form of energy that the body can use. The investigators propose that Gulf War Syndrome is determined by a complex interaction of factors that interfere with mitochondrial function. This study will be the first investigation of mitochondrial function in Gulf War Syndrome. The investigators objective is to establish the cause for symptoms in affected veterans, develop testing that can more easily identify Gulf War Syndrome, and ultimately develop treatment protocols for Gulf War Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Short-term memory loss or a severe inability to concentrate that affects work, school or other normal activities
* Muscle Pain, myalgias
* Pain without redness or swelling in a number of joints
* Intense or changing patterns of headaches
* Unrefreshing sleep
* After any exertion, weariness that lasts for more than a day

Exclusion Criteria:

* Organ failure (e.g. emphysema, cirrhosis, cardiac failure, chronic renal failure)
* Chronic infections (e.g. HIV/AIDS, hepatitis B or C)
* Rheumatic and chronic inflammatory diseases (e.g. systemic lupus erythematosis, Sjogren's syndrome, rheumatoid arthritis, inflammatory bowel disease, chronic pancreatitis.)
* Major neurologic diseases (e.g. multiple sclerosis, neuromuscular diseases, epilepsy or other disease requiring ongoing medication that could cause fatigue, stroke, head injury with residual neurologic deficits)
* Diseases requiring systemic treatment (e.g. organ or bone marrow transplantation; systemic chemotherapy; radiation of brain, thorax, abdomen, or pelvis)
* Major endocrine diseases (e.g. hypopituitarism, adrenal insufficiency)
* Myocardial infarction, heart failure
* Morbid obesity (body mass index >40)
* Permanent psychiatric exclusions: Lifetime diagnoses of bipolar affective disorders, schizophrenia or any subtype, delusional disorders of any subtype, dementias of any subtype, organic brain disorders, and alcohol or substance abuse within 2 years before onset of the fatiguing illness.
* History of allergic reaction to lidocaine
* History of keloid formation with skin incisions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gulf War Veterans who have been diagnosed with Gulf War Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Characterize mitochondrial cellular energetics in Gulf War Syndrome patients | approximately 2 years; once all data has been collected from study participants
  After collecting a skin and blood sample, mitochondrial cellular energetics in Gulf War Syndrome patients will be characterized by: 1. high resolution respirometry of intact cells, 2. quantitative analysis of individual mitochondrial proteins, 3. analysis of intact OXPHOS enzyme complexes and supercomplexes, 4. in gel enzyme activity assessment of intact OXPHOS enzyme complexes and supercomplexes, 5. mitochondrial DNA (mtDNA) copy number quantitation to assess for defects in regulation mtDNA replication and 6. cellular coenzyme Q10 quantitation.

SECONDARY OUTCOMES:
Mitochondrial DNA | approximately 2 years; once all data has been collected from study participants.
  Assess the mitochondrial DNA (mtDNA) from each patient with Gulf War Syndrome for mtDNA mutations by whole genome sequencing of leukocyte and skin cell mtDNA.

CONTACTS AND LOCATIONS:
Overall Officials: John M Shoffner, MD, Principal Investigator — Medical Neurogenetics
Locations (1):
- Medical Neurogenetics, LLC, Atlanta, Georgia, United States